CLINICAL TRIAL: NCT06955013
Title: Ability of Emergency Medicine Doctors to Use Ultrasound to View Muscle Layers of the Abdominal Wall
Brief Title: Ultrasound to View Abdominal Wall Muscle Layers
Status: Recruiting | Type: Observational
Sponsor: Corewell Health South (Other)
Responsible Party: Principal Investigator, Matthew Hysell, Medical Student Program Director, Corewell Health South
Other Study IDs: CHLIRB#1659
Record Dates: First submitted 2025-04-24; First posted 2025-05-02 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteers
Keywords: Ultrasound; Emergency Medicine; Abdominal Wall; Muscle Layers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy volunteer; BMI 29.9 and below
- Healthy volunteer; BMI 30 and above

SUMMARY:
The American College of Emergency Physicians (ACEP) views ultrasound-guided nerve blocks to be a core skill for emergency medicine physicians. They are used widely, commonly for various traumatic injuries, both for repair/stabilization of injuries, as well as for pain control while awaiting definitive management. Ultrasound is often used to identify specific nerves or fascial planes to guide deposition of local anesthetic. Some of these blocks include interscalene brachial plexus blocks to help manage shoulder dislocation, supraclavicular brachial plexus nerve blocks to help manage elbow dislocation or distal wrist fracture reductions, fascia iliaca plane block for pain control of hip fractures patients awaiting definitive surgery, and serratus anterior plane block to help manage rib fracture pain. As these techniques become more mainstream due to increasing focus upon them in residency training and improvements in ultrasound technology, research upon these blocks has increased dramatically since 2016, with most of these articles focusing on hip fracture and shoulder dislocation.

The abdominal musculature of the flank is comprised of the external oblique muscle, internal oblique muscle, and the transversus abdominis. Branches of the lateral cutaneous nerve pass between the internal oblique muscle innervating the peritoneum. First described in the anesthesia literature in 2001, transversus abdominis plane (TAP) block has been found to decrease narcotic requirement after abdominal surgery by targeting these branches. It has also been found to be effective when performed by surgeons. However, it has been only minimally alluded to in the emergency medicine literature.

Obesity can have a negative effect on image procurement in ultrasound. Given how little TAP blocks have been reviewed in the emergency medicine literature, even less is known about emergency physicians' ability to deal with added difficulties brought by increases in body habitus. Some anesthesia teachers recommend out-of-plane needle approaches in obese patients rather than in-plane needle approaches for less challenging body habituses. Ultrasound-guided TAP blocks have been used successfully in bariatric surgery, so there is precedent for use in this population.

The study proposes to evaluate emergency medicine physician ability to obtain images suitable for potential TAP block administration in patients with varying body habitus. The hypothesis is that while potential TAP block could be limited by increased body habitus, the majority of patients would still be able to potentially undergo the procedure.

Methods Approval for this study will be sought from the Lakeland IRB. This is a prospective study conducted at an academic community emergency department with a volume of about 69,000 annually. Patients were approached by emergency medicine residents on their ultrasound rotation with regards to willingness to participate in the study and written informed consent was obtained. Inclusion criteria were adult patients aged 18 and over who were willing to undergo the informal ultrasound looking to identify the muscular layers with enough definition that a TAP block could be carried out. No injection of medication was carried out in this study. Exclusion criteria included pediatric patients, patients unable to sign consent for themselves (including non-English speakers, patients with dementia or altered mental status), as well as populations potentially at risk (such as pregnant patients, prisoners, and minors). Patients with infectious considerations were excluded (such as those under isolation precautions or with open wounds/skin injury in the abdominal/flank area).

If patients were willing to participate, residents assigned patients a study number and recorded basic demographic information (age, sex, race, ethnicity, and Body Mass Index (BMI)). Residents then carried out the ultrasound starting with the linear array probe at the level of the umbilicus, fanning laterally to identify the rectus sheath and then the shared aponeurosis for the internal oblique and transversus abdominis muscle. The resulting image of the abdominal wall was then recorded, saved under the patient's study identification number, and saved digitally to the study folder maintained on hospital servers. Patients were only enrolled once. Patients were analyzed for differences in the rates of obtaining adequate images based on body habitus.

ELIGIBILITY:
Inclusion Criteria:

* Age: Adult patients aged 18 and over
* Willingness to participate: Patients who are willing to undergo the ultrasound procedure and provide written informed consent

Exclusion Criteria:

* Age: Pediatric patients (under 18 years old)
* Consent: Patients unable to sign consent for themselves, including non-English speakers, patients with dementia or altered mental status
* At-Risk Populations: Pregnant patients, prisoners, and minors
* Infectious Considerations: Patients under isolation precautions or with open wounds/skin injury in the abdominal/flank area

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients aged 18 and over who visit an academic community emergency department (ED) with an annual volume of approximately 69,000 patients. These patients are approached by emergency medicine residents during their ultrasound rotation and are asked to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 118 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Rates of success in obtaining adequate images | Up to one week after ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Hysell, Principal Investigator — Corewell Health South
Locations (1):
- Corewell Health Lakeland, Saint Joseph, Michigan, United States

IPD SHARING:
Plan to Share IPD: No